CLINICAL TRIAL: NCT01110122
Title: The Effect of Post-exercise Supplementation With Whey Protein Versus Carbohydrate on Soccer Performance.
Brief Title: Effect of Whey Protein on Soccer Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Ingeborg A Brouwer, VU University of Amsterdam
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AJA-PROT-IAB-001
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-03

CONDITIONS: Muscle Damage
Keywords: Muscle recovery; Intermittent exercise; Whey protein; Soccer
MeSH Terms: interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Whey protein — 20g, oral, dissolved in yoghurt-drink, after every training and match for 2 weeks

SUMMARY:
Rationale: During exercise protein breakdown in muscles is larger than protein synthesis. This negative muscle protein balance leads to increased muscle damage and thereby to a reduced muscle tissue recovery. To achieve a positive muscle protein balance and reduce muscle damage, many athletes use proteins. In professional soccer players, considerable stress is placed on the musculoskeletal system. Recovery time is often too short for these players to restore homeostasis, which results in catabolic processes. This increases playing errors and will lead to lapses in concentration. Therefore, it is of great importance for a professional soccer team to be in optimal condition and a fast recovery after exercise is desirable to accomplish maximum performance. Supplementation with whey proteins is thought to support this.

Objective: To assess whether post-exercise supplementation with whey protein will lead to a better muscle recovery than supplementation with carbohydrates in Dutch soccer players between the age of 15 and 18 years old.

Study design: A double blind randomised controlled cross-over trial.

Study population: Healthy soccer players of the A and B selection of AJAX between the age of 15 and 18 years old.

Intervention: Supplement, containing either whey proteins or an isocaloric carbohydrate placebo. Each supplement will be administered for 2 weeks separated by a 7 day washout period. Treatment order will be randomly assigned.

Main study parameters: The main study parameter will be the Yo-Yo intermittent recovery test level 2 score and the vertical jump test. The scores will evaluate the soccer players' ability to repeatedly perform intense exercise and his potential to recover from this exercise.

ELIGIBILITY:
Inclusion Criteria:

* performing soccer >1 year
* part of A & B selection of AJAX

Exclusion Criteria:

* presence of lactose intolerance
* presence of illness
* presence of injury

Ages: 15 Years to 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Muscle recovery | 2 weeks
  Recovery will be measured with the test scores on the Yo-Yo Intermittent Recovery Test level 2 and the Countermovement Jumping Test.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg A Brouwer, PhD, Principal Investigator — VU University of Amsterdam
Locations (1):
- Ajax, Amsterdam, Netherlands